CLINICAL TRIAL: NCT01694745
Title: European Survey of Sedation and Analgesia Practices for Newborns Admitted to Intensive Care Units
Brief Title: EUROpean Pain Audit In Neonates
Acronym: EUROPAINsurvey
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, CARBAJAL, Professor, Hôpital Armand Trousseau
Other Study IDs: EUROPAIN Survey
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2013-02

CONDITIONS: Pain; Analgesia; Sedation; Intesive Care; Intratracheal Ventilation
Keywords: Newborns; Premature; Pain; Pain assessment; Endotracheal Intubation; Analgesia; Sedation; Longterm effects of pain; Epidemiology
MeSH Terms: conditions — Pain; Agnosia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EUROPAIN Survey is an epidemiological study aimed at assessing current clinical practices regarding the use of sedative and analgesic drugs in newborns admitted to NICUs or PICUs in different countries in Europe. This study is conducted as part of the NeoOpiod study.

The main objective of this study is to determine the current clinical practices regarding the use of sedative and analgesic drugs in newborns in intensive units in different countries in Europe. The principal criteria are: the frequency of ventilated neonates receiving sedation and analgesia, the medications used for sedation and analgesia in ventilated neonates, the length of use of medications administered for sedation and analgesia in ventilated neonates and similarities and differences in sedation and analgesia practices among European countries.

The secondary objectives are: a) to determine the proportion of neonatal units that have developed and implemented local written guidelines to provide continuous sedation and analgesia in ventilated newborn infants as well as to prevent and treat procedural pain, b) to document the published guidelines for neonatal analgesia and sedation in different European countries and develop consensus for common European standards that can be applied in all medical settings, c) to determine the frequency of use of pain assessment tools in ventilated newborn infants and evaluate their impact on pain management practices and d) to determine practices to assess and prevent withdrawal syndromes.

The EUROPAIN STUDY is observational and therefore it will not interfere with routine practices of participating units. No changes in diagnostic, therapeutic or any managing strategy of patients are imposed by the participation in this study. This epidemiological study will only collect data on clinical practices in each unit. It will include all neonates up to a corrected age of 44 weeks post conception.

The maximum duration of data collection for every included infant is 28 days. Data collection will stop before 28 days if the infant leaves the unit (discharge, death, transfer to another hospital). Data will be entered on a secure web-based questionnaire.

DETAILED DESCRIPTION:
1.1 Background and rationale The alleviation of pain is a basic and human right regardless of age. Neonates do feel pain and it has been shown that preterm infants are even more vulnerable to pain than older infants. The more vulnerable preterm neonates are precisely those that are more exposed to pain. Neonates admitted to intensive care units, both neonatal intensive care unit (NICU) and pediatric intensive care unit (PICU), undergo dozens or even hundreds of painful procedures during their stay. These painful procedures include, for many of the ICU neonates, a tracheal intubation followed by mechanical ventilation. The pain and stress that are induced by mechanical ventilation as well as by repetitive procedures or painful diseases has led medical staff to use sedation and analgesia in neonates admitted to intensive care units. The subjectivity and difficulty inherent to pain measurement in neonates have probably contributed to a wide variety of neonatal sedation and analgesia practices. To date, these practices have been rarely studied.

Why would sedation and analgesia be necessary? Mechanical ventilation is a potentially painful intervention. Adults often describe mechanical ventilation as a painful and anxiety-provoking experience. The main objectives of sedation and analgesia are: reduction of pain, stress and irritability, promotion of blood pressure stability, promotion of ventilator synchrony and improvement of oxygenation. In the long term, reduced stress, as well as reduced fluctuations in oxygenation and blood pressure is believed to minimize the risks of neurological injury and death. However, the use of sedation and analgesia is only conceivable in the respect of the principle that must accompany all medical actions: first, do no harm.

Pain and stress undergone during the neonatal period can have deleterious short-term and long-term consequences. Some of these consequences have been reduced with adequate analgesic treatment. Current data show the necessity to give adequate sedation and analgesia to ventilated neonates.

Statements promoting the use of sedation and analgesia The increased awareness that neonates feel pain, the ethical obligation to treat this pain with analgesics, the growing body of evidence demonstrating that untreated neonatal pain can lead to altered reactivity to pain that persists throughout infancy and childhood as well as the need for a humane management of neonates have lead to the development of International and National Guidelines promoting the use of analgesics in the neonatal population. These Guidelines state that units that provide neonatal care should develop and implement guidelines concerning neonatal pain. However, the existing literature is still conflicting regarding the use of sedation and analgesia for ventilated neonates. Current data indicate that there is insufficient evidence to recommend the routine use of opioids in mechanically ventilated newborns and that opioids should be used selectively. Sedation and analgesia in non ventilated babies is extremely rare.

Practices across Europe and USA Data on sedation and analgesia practices in ventilated neonates are very rare. In 1995 the SOPAIN study carried out in the United States showed that factors predicting the use of on-going analgesia and sedation in neonates included: mechanical ventilation, higher gestational age, and male gender. In 2005, the French EPIPPAIN study showed that the rate of continuous sedation and analgesia was 69.6% in ventilated neonates with large variations among centers (16.7% to 90.9%). The most frequently used drugs were midazolam and morphine.

To date, there are no data permitting the comparison of neonatal pain management within the European countries. The availability of these data will enable comparison of practices with state-of-the-art knowledge.

Study Hypothesis

The EUROPAIN study is an epidemiological study that is based on the following hypothesis:

* Most newborn ventilated infants receive continuous sedation and analgesia.
* Non ventilated babies are not sedated.
* Morphine, fentanyl and midazolam are the most frequently drugs used in this setting.
* Infrequent use of validated pain assessment tools to monitor sedation and analgesia occurs in ventilated newborn infants.
* Most units have developed written local guidelines for sedation and analgesia in ventilated neonates, but huge variability exists among practitioners in the same unit, across different units in the same country, and across different countries in Europe.
* Development, dissemination, and regular updates of common European standards will improve the care and clinical outcomes of ventilated newborn infants.

1.2 Main objective • To determine the current clinical practices regarding the use of sedative and analgesic drugs for ventilated newborns in different countries in Europe.

1.3 Principal criteria

* The frequency of ventilated neonates receiving sedation and analgesia in different European units
* The medications used for sedation and analgesia in ventilated neonates across Europe.
* The length of use of medications administered for sedation and analgesia in ventilated neonates
* Similarities and differences in sedation and analgesia practices among European countries

1.4 Secondary objectives and criteria

* To determine the proportion of neonatal units that have developed and implemented local written guidelines to provide continuous sedation and analgesia in ventilated newborn infants as well as to prevent and treat procedural pain.
* To document the published guidelines for neonatal analgesia and sedation in different European countries and develop consensus for common European standards that can be applied in all medical settings.
* To determine the frequency of use of pain assessment tools in ventilated newborn infants and evaluate their impact on pain management practices.
* To determine practices to assess and prevent withdrawal syndromes. Secondary criteria
* Variations across European countries of the proportions of units that have developed and implemented local written guidelines for sedation and analgesia in ventilated neonates
* Identification and description of national guidelines for sedation and analgesia in neonates in all participating countries. Identification of recommended drugs.

1.5 Type of study

• Epidemiological observational study.

1.6 Study plan The EUROPAIN STUDY is observational and therefore it will not interfere with routine practices of participating units. No changes in diagnostic, therapeutic or any managing strategy of patients are imposed by the participation in this study. This epidemiological study will only collect data on clinical practices in each unit.

The inclusion criteria are:

• All neonates up to a corrected age of 44 weeks post conception. That means, for example, that a baby of 40 weeks gestational age can be included up to 28 days (4 weeks) of post natal age or that a baby of 32 weeks gestational age can be included up to 12 weeks of post natal age.

At the unit level

* No modifications of current managing protocols or strategies are required by the participation in the EUROPAIN STUDY. The unit coordinators will only provide data on local protocols to manage procedural pain and sedation and analgesia in neonates as well as on general statistics of the unit. All treatments are authorized for included neonates since this study does not include any intervention
* A nurse and physician coordinator as well as a data quality manager will be designated for each unit.

At the national level

• The country coordinator will provide data on national guidelines to treat or prevent procedural or continuous pain in neonates.

Data collection

* The duration of data collection for every included infant is 28 days. However, data collection will stop before 28 days if the infant leaves the unit (discharge, death, transfer to another hospital).
* Data will be collected on individual data collection forms. These forms include demographic data, modes of respiration, continuous or intermittent sedative, analgesic or neuro-blocking drugs, pain assessment and drug withdrawal practices.
* Paper patient data collection forms are written in English with a subtitled translation in the country language. The web-based databases display questionnaires in the country language.
* The data collection forms will be completed by the unit nurse or physician coordinator or the person that they will designate.
* For each center, the duration of the inclusion period will be one month.
* Data will be entered on a secure web-based questionnaire.

1.7 Justification of number of patients Regarding the number of neonates to include in order to show possible differences in sedation and analgesia practices among the participating European countries, we have considered a scenario where differences are small. Thus, we have chosen an effect size (W) of 0.1. We have also assumed that 15 countries will participate. Using NCSS-PASS 2008 software, we have found that a total sample size of 2303 neonates will achieve 90% power to detect an effect size (W) of 0.1 using a 14 degrees (15 centers) of freedom Chi-Square test with a significance level (alpha) of 0.05. Therefore, we aim at including an average of 154 neonates per participating country.

1.8 Main Actions carried out during the study

* In each country, the National Principal Investigators (NPI) will send invitations to join the study to all level 3 neonatal units of the country. The NPI will then communicate the names, emails and telephone numbers of the units that accept to participate to the EUROPAIN STUDY principal investigators
* The NPI is responsible for the coordination of all units in the country and ensures communication with the EUROPAIN STUDY principal investigators
* The NPI will collect demographic data about the participating country.
* A nurse and physician coordinator as well as a data quality manager will be designated for each unit. The nurse and physician coordinator are responsible for informing all the unit staff about the study.
* The EUROPAIN STUDY principal investigators have prepared a specifically designed web-based database to enter data. Data can be entered directly from the patient's file. A paper copy of this database will be distributed to allow centers that prefer to perform a preliminary entry on paper forms before entering data on the web-based database. The medical coordinator or a person that he (she) will choose will enter the data into these specifically designed databases.
* The physician coordinator will report general statistics of the unit such as number of beds, number of admission, year ventilator-days etc to the Europain study principal investigators.
* Every unit will also report existing local guidelines on sedation and analgesia in ventilated infants, including routines for withdrawal and on the use of pain assessment tools.
* MONITORING PANEL. A monitoring panel will be created to monitor the progress of the study. This panel will ensure communication with all the participating units. This monitoring panel will be constituted by two persons working full-time during the study period. They will be stationed in Paris and working under the responsibility of EUROPAIN STUDY principal investigators.

ELIGIBILITY:
Inclusion Criteria:

* • All neonates up to a corrected age of 44 weeks post conceptional. That means, for example, that an infant born at 40 weeks gestational age can be included up to 28 days (4 weeks) of post natal age or that a baby of 32 weeks gestational age can be included up to 12 weeks of post natal age.

NOTE: Since this is an observational epidemiological study, all eligible infants of the unit during the study period should be included.

Exclusion Criteria:

* • The only exclusion criteria of this observational study is the participation of the neonate in a research study including a randomization for the use of sedative or analgesic drugs in ventilated neonates.

Max Age: 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * All neonates up to a corrected age of 44 weeks post conception. That means, for example, that a baby of 40 weeks gestational age can be included up to 28 days (4 weeks) of post natal age or that a baby of 32 weeks gestational age can be included up to 12 weeks of post natal age.
  * The aim of including all neonates is to both ensure a generalization of the findings to all ventilated and non ventilated neonates admitted to intensive care units and to obtain a clear description of practices across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 6489 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The frequency of ventilated neonates receiving sedation and analgesia in different European units | one year

SECONDARY OUTCOMES:
The medications used for sedation and analgesia in ventilated neonates across Europe | one year
The length of use of medications administered for sedation and analgesia in ventilated neonates | one year
Similarities and differences in sedation and analgesia practices among European countries | one year

OTHER OUTCOMES:
Variations across European countries of the proportions of units that have developed and implemented local written guidelines for sedation and analgesia in ventilated neonates | one year
Identification and description of national guidelines for sedation and analgesia in neonates in all participating countries. Identification of recommended drugs | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carbajal, MD PhD, Principal Investigator — Armand Trousseau
Locations (242):
- Austria (4):
  - Universitäts-klinik für Kinder- und Jugendheilkunde Innsbruck, Innsbruck
  - Landeskran- kenhaus Leoben, Leoben
  - Universitäts-klinik für Kinder und Jugendheilkunde Salzburg, Salzburg
  - Universitäts klinik für Kinder-und Jugenheilkunde Wien, Vienna
- Belgium (4):
  - Universitaire Ziekenhuis Antwerpen, Antwerp
  - Hôpital Erasme ULB,, Brussels
  - Centre Hospitalier Universitaire Tivoli, La Louvière
  - Centre Hospitalier Régional de la Citadelle, Liège
- Neonatal Intensiv Care Unit, Arch. Makarios Hospital, Nicosia, Cyprus
- Estonia (2):
  - Department of Anesthesiology and Intensive Care, Tallinn Children's Hospital, Tallinn
  - Paediatric Intensive Care Unit, Clinic of Anaesthesiology and Intensive Care, Tartu University Clinics, Tartu
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (34):
  - CHR Félix Guyon, Saint-Denis, La Réunion
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Arras, Arras
  - CH Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU Caen, Caen
  - CH Chambéry, Chambéry
  - CH Cherbourg, Cherbourg
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CH Le Havre, Le Havre
  - CH Le Mans, Le Mans
  - CHU Lyon Croix Rousse, Lyon
  - Hôpital Femme,Mère, enfant, Lyon
  - Hôpital de la conception - APHM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - CHU de Nîmes, Nîmes
  - CHR Orléans, Orléans
  - CHU Pau, Pau
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CH Rouen, Rouen
  - Ch Saint Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CH Troyes, Troyes
  - CH Bretagne Atlantique, Vannes
- Germany (4):
  - Klinik fUr Kinder und Jugendliche Sozialstiftung Bamberg, Bamberg
  - Klinikum Coburg, Coburg
  - Department of Paediatric and Adolescent Medicine University Hospital Erlangen, Erlangen
  - Cnopf'sche Kinderklinik, Nuremberg
- Greece (13):
  - "Gaia" Maternity Hospital, Athens
  - "Lito" Maternity Hospital, Athens
  - "Mitera" General Maternity and Pediatric Clinic, Athens
  - "Rea" Maternity Hospital, Athens
  - Alexandras Hospital general, Athens
  - Children's Hospital "Agia Sophia", Athens
  - Helena Venilezoy Maternit y Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University of Ioannina, Ioannina
  - University of Patras, Pátrai
  - 1st Dept of Neonatalogy, Aristole University of Thessaloniki, Thessaloniki
  - 2nd Dept of Neonatalogy, Aristole University of Thessaloniki, Thessaloniki
  - Menn Esy, Hippokratio General Hospital, Thessaloniki
- Italy (28):
  - TIN Ospedale San Giovanni di Dio, Agrigento
  - UO TIN Neonatologia AOU Sant'Orsola Malpighi, Bologna
  - TIN Bolzano, Bolzano
  - UO TIN e Patologia Neonatale, Camposampiero
  - TIN Como Valduce, Como
  - U.O. di Neonatologia e PatNeo con T.I. - Istituti Ospitalieri, Cremona
  - Ospedale Careggi, Florence
  - Patologia Neonatale Lodi, Lodi
  - IN Ospedale Macedonio Melloni Milano-AO Fatebenefratellied Oftalmico, Milan
  - TIN Centro IRCSS Ca Granda-Policlinico Osp.Maggiore Mangiagalli LI, Milan
  - TIN Modena, Modena
  - TIN/Neonatologia- fondazione MBBM- H San Gerardo, Monza
  - TIN E Patologia Neonatale Dip. di Salute della donna e del bambino- Università di Padova, Padua
  - UTIN Perugia, Perugia
  - UO Neonatologia Santa Chiara, Pisa
  - TIN A.O.Bianchi-Melacrino-Morelli, Reggio Calabria
  - Azienda Ospedaliera ASMN, Reggio Emilia, Reggio Emilia
  - NICU Rimini, Rimini
  - TIN Ospedale Pediatrico Bambino Gesù, Roma
  - TIN Ospedale San Pietro FBF, Roma
  - Azienda Ospedaliera Universitaria di Sassari, Sassari
  - Ospedale Maria Vittoria, Torino, Torino
  - UO Neonatologia e TIN Ospedale Santa Chiara, Trento
  - UO TIN e Patologia Neonatale, Treviso
  - Patologia Neonatale Ospedale S.M.Misericordia, Udine
  - Terapia Intensiva Neonatale e Pediatrica, Verona
  - U.O.Patologia e Terapia Intensiva Neonatale AOUI Borgo Roma, Verona
  - TIN Ospedale San Bortolo, Vicenza
- Department of Neonatology Lithuanian University of Health Sciences,, Kaunas, Lithuania
- Mater Dei Hospital, Triq Dun Karm, Msida, Malta
- Netherlands (5):
  - Academic medical Center Amsterdam - Emma Children's Hospital, Amsterdam
  - ErasmusMC - Sophia Childrens Hospital, Rotterdam
  - University Hospital Utrecht - Wilhelmina Children's Hospital, Utrecht
  - Maxima Medical Center Veldhoven, Veldhoven
  - Isala Clinics Zwolle - Amalia Children's Hospital, Zwolle
- Norway (16):
  - Aalesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordland Hospital, Bodø
  - Vestre Viken Hospital, Drammen
  - Ostfold Hospital, Fredrikstad
  - Haugesund Hospital, Haugesund
  - Sorlandet Hospital, Kristiansand
  - Sykehuset Innlandet Lillehammer, Lillehammer
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital - Rikshospitalet, Oslo
  - Oslo University Hospital - Ullevaal, Oslo
  - Telemark Hospital, Skien
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs hospital, Trondheim
  - Vestfold Hospital, Tønsberg
- Poland (8):
  - Oddzial Noworodkow, Bydgoszcz
  - Szpital Wojewódzki Koszalin, Koszalin
  - Children's Memorial Health Institute Warsaw, Warsaw
  - Clinical Hospital Ks.Anna Mazowiecka, Warsaw
  - Department of obstetric and gynecology, medical University of Warsaw, Warsaw
  - Hospital Orłowskiego Warsaw, Warsaw
  - Oddział Neonatologiczny, Warsaw
  - Departement of Neonato- logy Medical University in Wrocław, Wroclaw
- Portugal (14):
  - Hospitale Divino Espirito Santo, Açores
  - Hospital San Marcos, Braga
  - Maternidade Bissaya Barreto, Coimbra
  - Maternidade Daniel Matos, Coimbra
  - Hospitale Espirito Santa, Evora
  - Hospitale Faro, Faro
  - Hospitale Vila Nova Gaia, Gaia
  - Hospital Dona Estefânia, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospitale Amadora Sintra, Lisbon
  - Hospitale Sao Francisco Xavier, Lisbon
  - Maternity Dr Alfredo da Costa, Lisbon
  - Hospitale Funchal, Madeirã
  - Hospital San João, Porto
- Spain (30):
  - Complexo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario Principe de Asturias, Alcalá de Henares
  - Hospital General de Alicante, Alicante
  - Hospital Universitario de Álava, Álava
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General de Castellón, Castellon
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitari Josep Trueta, Girona
  - Hospital Universitario Severo Ochoa, Leganés. Madrid
  - Hospital San Pedro de Logroño, Logroño
  - Hospital Clínico San Carlos (Madrid), Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Complexo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen de la Salud (Toledo), Toledo
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Complexo Hospitalario Universitario de Vigo, Vigo
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (6):
  - Hospital Lasarettet, Falun
  - Universitetssjukhuset, Lund
  - Universitetssjukhuset, Örebro
  - Karolinska University Hospital (Stockholm), Stockholm
  - Sachsska Barnsjukhuset (Stockholm), Stockholm
  - Akademiska Barnsjukhuset, Uppsala
- United Kingdom (66):
  - Aberdeen Maternity Hospital, Aberdeen
  - Royal United Hospital, Bath
  - Royal Berkshire NHSFT, Berkshire
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Birmingham Womens Hospital, Birmingham
  - Sandwell and West Birmingham, Birmingham
  - Blackpool Teaching Hospital Foundation Trust, Blackpool
  - Royal Bolton Hospital, Bolton
  - Bradford Royal Infirmary, Bradford
  - Royal Alexander Children's Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - Southmead Hospital, Bristol
  - St Michael's Hospital, Bristol NICU, Bristol
  - Royal Brompton Hospital, Brompton
  - Burnley General Hospital, Burnley
  - Countess of Chester, Chester
  - North Tees Hospital, Cleveland
  - Colchester General Hospital, Colchester
  - University Hospitals Coventry & Warwick, Coventry
  - Royal Derby Hospital, Derby
  - Royal Devon and Exeter NHS Foundation Trust, Devon
  - Doncaster Royal Infirmary, Doncaster
  - Edinburgh Royal Infirmary, Edinburgh
  - Medway Maritime Hospital, Gillingham
  - Gloucestershire Royal Hospital, Gloucestershire
  - Royal Gwent Hospital, Gwent
  - Airedale NHS Foundation Trust, Keighley
  - Kettering General Hospital, Kettering
  - Leeds General Infirmary, Leeds
  - Leicester Royal infirmary NICU, Leicester
  - Leicester Royal Infirmary PICU, Leicester
  - Leighton or Mid Cheshire NHS Trust, Leighton
  - Liverpool Women's Hospital NICU, Liverpool
  - Evelina Children's Hospital, Guy's and St Thomas' NHS Foundation Trust PICU, London
  - Great Ormond Street Hospital for Sick Children PICU, London
  - Imperial College London NICU, London
  - Royal London Hospital, London
  - Pennine Acute Hospitals NHS Trust, Manchester
  - St Mary's Hospital, Manchester
  - King's Mill Hospital, Mansfield, Mansfield
  - James Cook University Hospital, Middlesborough, Middlesbrough
  - West Middlesex University Hospital, Middlesex
  - Newham University Hospital, Newham
  - Northampton General Hospital Neonatal Unit, Northampton
  - Queen's Medical Centre, Nottingham
  - Southport & Ormskirk & District General Hospital Neonatal Unit, Ormskirk
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth, Plymouth
  - Royal Preston Hospital, Preston
  - Queen's Hospital, Romford, Romford
  - Rotherham District General Hospital, Rotherham
  - Jessop Wing, Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - Singleton Hospital, Singleton
  - University Hospital Of North Staffordshire NHS Trust, Staffordshire
  - Great Western Hospitals NHS Foundation Trust, Swindon
  - Musgrove Park Hospital, Taunton, Taunton
  - Royal Cornwall Hospital, Treliske
  - Warrington Hospital, Warrington
  - Calderdale Royal Hospital, West Yorkshire
  - Pinderfields General Hospital, West Yorkshire
  - New Cross Hospital, Wolverhampton, Wolverhampton
  - Worcester Royal Hospital, Worcester
  - University Hospital of South Manchester, Wythenshawe, Wythenshawe
  - York Teaching Hospital NHS Foundation Trust, York

REFERENCES:
- [Derived] Lago P, Frigo AC, Baraldi E, Pozzato R, Courtois E, Rambaud J, Anand KJ, Carbajal R. Sedation and analgesia practices at Italian neonatal intensive care units: results from the EUROPAIN study. Ital J Pediatr. 2017 Mar 7;43(1):26. doi: 10.1186/s13052-017-0343-2. PMID 28270167
- [Derived] Carbajal R, Eriksson M, Courtois E, Boyle E, Avila-Alvarez A, Andersen RD, Sarafidis K, Polkki T, Matos C, Lago P, Papadouri T, Montalto SA, Ilmoja ML, Simons S, Tameliene R, van Overmeire B, Berger A, Dobrzanska A, Schroth M, Bergqvist L, Lagercrantz H, Anand KJ; EUROPAIN Survey Working Group. Sedation and analgesia practices in neonatal intensive care units (EUROPAIN): results from a prospective cohort study. Lancet Respir Med. 2015 Oct;3(10):796-812. doi: 10.1016/S2213-2600(15)00331-8. Epub 2015 Sep 24. PMID 26420017
- See also: Study website — http://www.europainsurvey.eu